CLINICAL TRIAL: NCT04319328
Title: Pharmacokinetic Evaluation of Cefazolin, Ceftazidime, and Ciprofloxacin in Chronic Hemodialysis Patients
Brief Title: Is Cefazolin, Ceftazidime and Ciprofloxacin Dosing Optimal in Hemodialysis Patients?
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: The Kidney Foundation of Canada (Other)
Responsible Party: Principal Investigator, Sheryl Zelenitsky, Professor, College of Pharmacy, Rady Faculty of Health Sciences, University of Manitoba
Other Study IDs: H2019:031
Record Dates: First submitted 2020-03-02; First posted 2020-03-24 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Hemodialysis Complication; Infectious Disease; End Stage Renal Disease
Keywords: Hemodialysis; Pharmacokinetics; Antibiotic Dosing; Cefazolin; Ceftazidime; Ciprofloxacin
MeSH Terms: conditions — Communicable Diseases; Kidney Failure, Chronic | interventions — Cefazolin; Ceftazidime

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cefazolin: n = 20
  Interventions: Drug: Cefazolin
- Ceftazidime: n = 20
  Interventions: Drug: Ceftazidime
- Ciprofloxacin: n = 20

INTERVENTIONS:
Drug: Cefazolin — Non-interventional pharmacokinetic evaluation
  Groups: Cefazolin
Drug: Ceftazidime — Non-interventional pharmacokinetic evaluation
  Groups: Ceftazidime

SUMMARY:
This study aims to optimize the dosing of cefazolin, ceftazidime, and ciprofloxacin for patients on high-flux hemodialysis. For each antibiotic 20 participants will be enrolled and three blood samples will be collected from each participant. Antibiotic levels will be measured in each blood sample. This data will be used to develop population-pharmacokinetic models for each antibiotic. Finally, Monte Carlo simulations will be used to develop evidence-based dosing recommendations.

DETAILED DESCRIPTION:
The goal of this study is to optimize the dosing of three commonly used antibiotics, thereby improving the treatment of serious, often life-threatening infections in patients on intermittent high-flux hemodialysis (iHFHD).

The hypothesis is that current antibiotic dosing is suboptimal, thereby increasing the risk of poor outcomes including treatment failure, adverse drug reactions and antibiotic resistance.

A prospective, non-interventional pharmacokinetic (PK) study of cefazolin, ceftazidime, and ciprofloxacin will be conducted in the St. Boniface Hospital outpatient hemodialysis unit.

The 1st objective of this study is to measure the free and total plasma concentrations of cefazolin, ceftazidime, and ciprofloxacin in adult patients on iHFHD and receiving antibiotic therapy for suspected or proven infection. For each antibiotic 20 participants will be enrolled and three blood samples will be collected from each participant. Antibiotic concentrations will be measured using an ultra high performance liquid chromatograph mass spectrometer. Total antibiotic concentrations in plasma will be measured in all patient samples. To describe protein binding, free levels will also be measured in the first two samples collected from the first 10 patients for each antibiotic.

The 2nd objective of this study is to characterize the PK of cefazolin, ceftazidime, and ciprofloxacin in patients on iHFHD using population-PK modelling. Covariates with potential influence on PK such as gender, age, body weight, dialyzer type, blood and dialysate flow rates, duration of dialysis and Kt/Vurea will be investigated, and incorporated as appropriate. For each antibiotic, the best PK model will be selected using established goodness-of-fit tests, and then independently validated.

The 3rd objective of this study is to translate findings to patient care using Monte Carlo simulations to evaluate conventional antibiotic dosing and develop optimized evidence-based dosing recommendations for cefazolin, ceftazidime, and ciprofloxacin in patients on iHFHD.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Proven or suspected infection
* Receiving cefazolin, ceftazidime, or ciprofloxacin for treatment
* Treatment course allows for collection of three 6 mL blood samples as per protocol

Exclusion Criteria:

* Chronic liver disease, Child Pugh Class C or higher
* Received study drug as part of a different treatment course in 1-week preceding start of new treatment course
* Acute kidney injury or recovering kidney function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients on chronic intermittent high-flux hemodialysis being treated for infection.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Volume of distribution (Vd) for cefazolin, ceftazidime, and ciprofloxacin in infected patients on chronic intermittent high-flux hemodialysis. | 48 to 72 hours
Drug elimination (ke) for cefazolin, ceftazidime, and ciprofloxacin in infected patients on chronic intermittent high-flux hemodialysis. | 48 to 72 hours
  Drug elimination (ke) during and between dialysis sessions
Drug clearance (CL) for cefazolin, ceftazidime, and ciprofloxacin in infected patients on chronic intermittent high-flux hemodialysis. | 48 to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl A Zelenitsky, PharmD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - Saint Boniface Hospital, Outpatient Hemodialysis Unit, Winnipeg, Manitoba
  - College of Pharmacy, University of Manitoba, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: Undecided